CLINICAL TRIAL: NCT03161405
Title: A Single-Sequence, Open-Label, 2-Period, Crossover Trial to Evaluate the Effect of the Potent CYP3A4 Inhibitor Itraconazole on the Single-Dose Pharmacokinetics of Oral TAK-906 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of the Potent CYP3A4 Inhibitor Itraconazole on the Pharmacokinetics (PK) of TAK-906 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-906-1003; U1111-1192-7802 (Registry Identifier: WHO)
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-07

CONDITIONS: Healthy Participants
Keywords: Drug Therapy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-906 maleate 25mg;Itraconazole 200mg + TAK-906 maleate 25mg (Experimental): TAK-906 maleate 25 milligram (mg), capsule, orally, once on Day 1 of First Intervention Period, followed by a minimum of 4-day washout period, further followed by Itraconazole 200 mg, solution, orally, once daily on Days 1 to 5 along with TAK-906 maleate 25 mg, capsule, orally on Day 4 of Second Intervention Period.
  Interventions: Drug: TAK-906 Maleate; Drug: Itraconazole

INTERVENTIONS:
Drug: TAK-906 Maleate — TAK-906 capsule
Drug: Itraconazole — Itraconazole solution

SUMMARY:
The purpose of this study is to evaluate the effect of the potent cytochrome P-450 (CYP) 3A4 inhibitor (itraconazole) on the single-dose PK of oral TAK-906 maleate.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-906. TAK-906 is being tested in healthy participants in order to evaluate the effect of the potent CYP3A4 inhibitor itraconazole on the single-dose PK of TAK-906 maleate.

The study enrolled 12 participants. Participants received the following treatment sequence:

• TAK-906 maleate 25 mg; Itraconazole 200 mg + TAK-906 maleate 25 mg

Participants were given an oral dose of TAK-906 in the First Intervention Period which was followed by a washout period, after which participants were given Itraconazole solution along with TAK-906 orally in the Second Intervention Period.

This single center trial was conducted in the United States. The overall duration to participate in this study was 7 weeks. Participants remained confined in the clinic from Day 1 up to Day 2 (First Intervention Period) and Day 4 up Day 6 (Second Intervention Period). Participants returned for a Follow-up Visit, 10 to 14 days after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Is a man or woman (with no child bearing potential) aged 18 to 55 years, inclusive, at the Screening Visit.
2. Has a body mass index (BMI) greater than or equal to (>=) 18 and less than or equal to (<=) 30 kilogram per square meter (kg/m^2) and a body weight greater than (>) 50 kilogram (kg) at the Screening Visit.
3. Is a nonsmoker who has not used tobacco- or nicotine-containing products (example, nicotine patch) for at least 6 months before administration of the initial dose of trial drug/invasive procedure.

Exclusion Criteria:

1. Has a positive alcohol or drug screen.
2. Has had a major surgery, donated or lost 1 unit of blood (approximately 500 milliliter [mL]) within 8 weeks of the first dose of study drug.
3. Has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce] per day).
4. Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
5. Has a substance abuse disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-07-02 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Takeda Investigational Site, Lenexa, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 05 June 2017 to 10 July 2017.
Pre-assignment Details: Healthy participants were enrolled in single sequence 2-period crossover study to receive TAK-906 maleate 25 milligram (mg) in First Intervention Period followed by Itraconazole 200 mg along with TAK-906 maleate 25 mg in Second Intervention Period.
Groups:
- TAK-906 Maleate 25mg;Itraconazole 200mg + TAK-906 Maleate 25mg: TAK-906 maleate 25 mg, capsule, orally, once on Day 1 of First Intervention Period, followed by a minimum of 4-day washout period, further followed by Itraconazole 200 mg, solution, orally, once daily on Days 1 to 5 along with TAK-906 maleate 25 mg, capsule, orally on Day 4 of Second Intervention Period.
Period: First Intervention Period (3 Days)
Arm/Group | TAK-906 Maleate 25mg;Itraconazole 200mg + TAK-906 Maleate 25mg
Started | 12
Completed | 12
Not Completed | 0
Period: Washout Period (at Least 4 Days)
Arm/Group | TAK-906 Maleate 25mg;Itraconazole 200mg + TAK-906 Maleate 25mg
Started | 12
Completed | 12
Not Completed | 0
Period: Second Intervention Period (6 Days)
Arm/Group | TAK-906 Maleate 25mg;Itraconazole 200mg + TAK-906 Maleate 25mg
Started | 12
Completed | 11
Not Completed | 1
Not completed — Positive urine drug screen | 1

BASELINE CHARACTERISTICS:
Population: The safety set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | TAK-906 Maleate 25mg;Itraconazole 200mg + TAK-906 Maleate 25mg
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 85.4 (10.59)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 180.8 (6.79)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.2 (2.52)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-906
Time Frame: TAK-906 maleate 25mg: Day 1 pre-dose and at multiple time points (up to 48 hours) post-TAK-906 maleate-dose; Itraconazole 200 mg + TAK-906 maleate 25mg: Day 4 pre-dose and at multiple time points (up to 48 hours) post- TAK-906 maleate-dose
Population: The pharmacokinetic (PK) analysis set included all participants from the safety set who had at least 1 measurable post-dose TAK-906 plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- TAK-906 Maleate 25 mg: TAK-906 maleate 25 mg, capsule, orally, once on Day 1 of First Intervention Period.
- Itraconazole 200 mg + TAK-906 Maleate 25 mg: Itraconazole 200 mg, solution, orally, once daily on Days 1 to 5 along with TAK-906 maleate 25 mg, capsule, orally on Day 4 of Second Intervention Period.
Arm/Group | TAK-906 Maleate 25 mg | Itraconazole 200 mg + TAK-906 Maleate 25 mg
Number analyzed (Participants) | 12 | 11
nanogram per milliliter (ng/mL) | 9.532 (4.6337) | 17.999 (4.8780)
Statistical Analysis 1: Comparison: TAK-906 Maleate 25 mg vs Itraconazole 200 mg + TAK-906 Maleate 25 mg; A paired t-test on the natural log-transformed parameters was performed. The mean difference and its 90 percent (%) confidence interval (CI) for the log-transformed parameters were exponentiated to obtain the point estimates of the itraconazole effect and 90% CIs; Test type: Other; Geometric mean ratio = 1.9827, 90% CI 2-sided [1.6446 to 2.3904]

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-906
Time Frame: as for outcome 1
Population: The PK analysis set included all participants from the safety set who had at least 1 measurable post-dose TAK-906 plasma concentration.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | TAK-906 Maleate 25 mg | Itraconazole 200 mg + TAK-906 Maleate 25 mg
Number analyzed (Participants) | 12 | 11
hour*nanogram per milliliter (h*ng/mL) | 24.10 (8.173) | 30.73 (8.521)
Statistical Analysis 1: Comparison: TAK-906 Maleate 25 mg vs Itraconazole 200 mg + TAK-906 Maleate 25 mg; A paired t-test on the natural log-transformed parameters was performed. The mean difference and its 90% CI for the log-transformed parameters were exponentiated to obtain the point estimates of the itraconazole effect and 90% CIs; Test type: Other; Geometric mean ratio = 1.2914, 90% CI 2-sided [1.1199 to 1.4891]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-906
Time Frame: as for outcome 1
Population: The PK analysis set included all participants from the safety set who had at least 1 measurable post-dose TAK-906 plasma concentration. PK analysis set where Day 1 and 4 assessments were available.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TAK-906 Maleate 25 mg | Itraconazole 200 mg + TAK-906 Maleate 25 mg
Number analyzed (Participants) | 12 | 11
h*ng/mL | 24.41 (8.136) | 31.45 (8.995)
Statistical Analysis 1: Comparison: TAK-906 Maleate 25 mg vs Itraconazole 200 mg + TAK-906 Maleate 25 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Geometric mean ratio = 1.2783, 90% CI 2-sided [1.0965 to 1.4904]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose study drug up to 30 days after the last dose of study (approximately Day 36)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Itraconazole 200 mg: Itraconazole 200 mg, solution, orally, once daily on Days 1 to 3 of Second Intervention Period.
- Itraconazole 200 mg + TAK-906 Maleate 25 mg: Itraconazole 200 mg, solution, orally, once daily on Days 4 and 5 along with TAK-906 maleate 25 mg, capsule, orally on Day 4 of Second Intervention Period.
Arm/Group | TAK-906 Maleate 25 mg | Itraconazole 200 mg | Itraconazole 200 mg + TAK-906 Maleate 25 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 1/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-906 Maleate 25 mg (N=12) | Itraconazole 200 mg (N=11) | Itraconazole 200 mg + TAK-906 Maleate 25 mg (N=11)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT03161405/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT03161405/SAP_001.pdf